CLINICAL TRIAL: NCT03670069
Title: A Pilot Study Examining the Impact of the Jak1 Inhibitor Itacitinib on the Sarcoma Tumor Immune Microenvironment
Brief Title: Itacitinib in Treating Patients With Refractory Metastatic/Advanced Sarcomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated early with 27 out of 28 planned subjects enrolled. This decision was multifactorial, including slow enrollment in the last remaining cohort and a lack of evidence of clinical benefit.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG9218021; NCI-2018-00615 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9715 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Metastatic Leiomyosarcoma; Metastatic Synovial Sarcoma; Metastatic Undifferentiated Pleomorphic Sarcoma; Advanced Myxoid Liposarcoma; Advanced Soft Tissue Sarcoma; Metastatic Myxoid Liposarcoma; Metastatic Round Cell Liposarcoma; Metastatic Soft Tissue Sarcoma; Refractory Leiomyosarcoma; Refractory Myxoid Liposarcoma; Refractory Round Cell Liposarcoma; Refractory Soft Tissue Sarcoma; Refractory Synovial Sarcoma; Refractory Undifferentiated Pleomorphic Sarcoma; Advanced Leiomyosarcoma; Advanced Synovial Sarcoma; Advanced Undifferentiated Pleomorphic Sarcoma; Metastatic Chondrosarcoma
MeSH Terms: conditions — Leiomyosarcoma; Sarcoma, Synovial; Histiocytoma, Malignant Fibrous; Liposarcoma, Myxoid; Sarcoma; Chondrosarcoma | interventions — itacitinib; baricitinib; INCB039110

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (itacitinib) (Experimental): Patients receive itacitinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Itacitinib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Itacitinib — Given PO
  Other Names: 1334298-90-6; 3-Azetidineacetonitrile; INCB039110
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot phase I trial studies how well itacitinib works in treating patients with sarcomas that do not respond to treatment (refractory) and have spread to other parts of the body (advanced/metastatic). Itacitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive itacitinib orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 7 and 30 days, every 12 weeks from baseline for up to 1 year, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Subjects >= 18 years old
* Must have a histologically confirmed diagnosis of sarcoma with one of the following subtypes:

  * Cohort 1: Leiomyosarcoma
  * Cohort 2: Undifferentiated pleiomorphic sarcoma
  * Cohort 3: Synovial sarcoma or myxoid/round cell liposarcoma
  * Cohort 4: Chondrosarcoma (all subtypes of chondrosarcoma are allowed)
* Subjects enrolling to cohorts 1, 2, or 3 must have received at least two prior lines of systemic therapy. Subjects enrolling to cohort 4 only may have received any number of prior lines of systemic therapy or may be treatment naïve
* All ongoing toxicities related to prior therapies must be resolved to grade 1 or better (except alopecia)
* Subjects must have one or more measurable lesions, as determined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 assessed by computed tomography (CT) or magnetic resonance imaging (MRI)
* Subjects must have at least one superficial lesion accessible for multiple biopsies; the tumor being biopsied cannot have been previously targeted for radiation therapy or have previously received intra-lesional treatment

  * NOTE: Superficial lesions previously targeted with radiation therapy that have demonstrated significant new growth via radiological imaging may be targeted for biopsy, with sponsor-investigator approval.
* Total bilirubin level =< 1.5 x the upper limit of normal (ULN) range mg/dL
* Aspartate aminotransferase (AST) =< 2.5 x ULN and alanine aminotransferase (ALT) levels =< 2.5 x ULN
* Alkaline phosphatase < 2.5 x ULN
* Serum creatinine =< 1.5 x ULN
* Calculated creatinine clearance >= 30 mL/min using the Cockcroft-Gault formula may be included
* Absolute neutrophil count (ANC) >= 1.5 × 10^9/L
* Platelet count >= 100 x 10^9/L; transfusion is permitted as clinically indicated
* Hemoglobin >= 9 g/dL

  * Transfusion is permitted as clinically indicated
* Subjects must have a life expectancy >= 6 months, as determined by the treating physician
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 or Karnofksy performance status >= 60
* Male or non-pregnant and non-breast feeding female:

  * Females of child-bearing potential must agree to use highly effective contraception without interruption from initiation of therapy and while on study medication and have a negative serum pregnancy test (beta - human chorionic gonadotropin [hCG]) result at screening and agree to ongoing pregnancy testing during the course of the study, and at the end of study treatment; a highly effective method of contraception is defined as one that results in a low failure rate (that is, < 1% per year), when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine contraceptive devices, sexual abstinence, or a vasectomized partner
  * Male subjects must practice abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study
* Ability to understand and sign informed consent document
* Willingness and ability to comply with scheduled visits, laboratory tests, and other study procedures

Exclusion Criteria:

* Known active, uncontrolled, or symptomatic central nervous system (CNS) metastases; a subject with controlled and asymptomatic CNS metastases may participate in this study; as such, the subject must have completed any prior treatment for CNS metastases >= 28 days (including radiotherapy and/or surgery) prior to the start of treatment in this study and should not be receiving chronic corticosteroid therapy for CNS metastases; subjects with known CNS metastases must be confirmed radiographically stable by at least one imaging study, at least 28 days from last treatment
* Receipt of any type of cytotoxic, biologic, or other systemic anticancer therapy (including investigational) within 2 weeks of enrollment
* Prior treatment with a drug targeting JAK1, JAK1/2 or STAT3 inhibitor; Food and Drug Administration (FDA) approved small molecule tyrosine kinase inhibitors (TKIs) not specifically designed to target this pathway are okay (e.g. pazopanib, sunitinib, sorafenib)
* Known, active drug or alcohol abuse
* Pregnant or lactating females
* Active or recent infection requiring systemic anti-infective treatment that was completed =< 14 days prior to enrollment (with the exception of uncomplicated urinary tract infection or upper respiratory infection)
* Uncontrolled or concurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Oral steroid usage within =< 14 days prior to enrollment
* Known inflammatory or autoimmune disease which requires patient to occasionally require high dose oral steroids
* Subjects with known, active human immunodeficiency virus (HIV) infection (subjects with undetectable viral load and normal CD4+ T-cell count are permitted)
* Inability to swallow food or tablets, or significant gastrointestinal disorder that, in the opinion of the investigator, could interfere with absorption of the study drug
* Previous reaction to any component of itacitinib or known hypersensitivity to the active substance or any of the excipients
* Subjects with a sarcoma which has other, defined treatments or biology distinctly different from those of soft tissue sarcomas in general; including, but not limited to, Ewing's sarcoma, rhabdomyosarcoma, gastrointestinal stromal tumors, Kaposi's sarcoma, Wilm's tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Difference in the percentage of cells which are immune inhibitory (CD11B+, CD163+) macrophages from pre-treatment to first post-treatment biopsy | From baseline to 2 years
  Evaluation of the change in percentages of cells against the null hypothesis of no difference will be performed using a 1-sided t-test at the 0.05 level.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 2 years
  Will be graded according to Common Terminology Criteria for Adverse Events version 5.0. The frequency and severity of toxicities will be evaluated by proportions and associated 95% confidence intervals.
Progression-free survival rate | At 6 months
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Distributions and percentages at landmark times for time to event outcomes will be estimated using the method of Kaplan-Meier. Confidence intervals about medians will be estimated using the method of Brookmeyer-Crowley. With 12 LMS patients, binary proportions can be estimated to within 29% with 95% confidence. With 8 (SS or MRCL) and PUS, respectively, binary proportions can be estimated to within 36% with 95% confidence.
Median overall survival | At 12 months
  Distributions and percentages at landmark times for time to event outcomes will be estimated using the method of Kaplan-Meier. Confidence intervals about medians will be estimated using the method of Brookmeyer-Crowley. With 12 LMS patients, binary proportions can be estimated to within 29% with 95% confidence. With 8 (SS or MRCL) and PUS, respectively, binary proportions can be estimated to within 36% with 95% confidence.
Clinical benefit rate (complete response [CR]+ partial response [PR]+stable disease [SD]) | At 12 weeks
  CR and PR will be defined as per RECIST 1.1 Distributions and percentages at landmark times for time to event outcomes will be estimated using the method of Kaplan-Meier. Confidence intervals about medians will be estimated using the method of Brookmeyer-Crowley. With 12 LMS patients, binary proportions can be estimated to within 29% with 95% confidence. With 8 (SS or MRCL) and PUS, respectively, binary proportions can be estimated to within 36% with 95% confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Cranmer, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/69/NCT03670069/ICF_000.pdf